CLINICAL TRIAL: NCT01200992
Title: A Phase 3, Randomized, Active-Controlled, Open-Label, Multicenter Study to Evaluate the Efficacy and Safety of EN3348 (MCC) as Compared With Mitomycin C in the Intravesical Treatment of Subjects With BCG Recurrent or Refractory Non-Muscle Invasive Bladder Cancer
Brief Title: Efficacy and Safety Evaluation of EN3348 (Mycobacterial Cell Wall-DNA Complex [MCC]) as Compared With Mitomycin C in the Intravesical Treatment of Subjects With BCG Recurrent/Refractory Non-muscle Invasive Bladder Cancer
Acronym: EMBARC-RF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of Recruitment
Sponsor: Bioniche Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EN3348-303
Record Dates: First submitted 2010-09-12; First posted 2010-09-14 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Bladder Neoplasm; Neoplasm Recurrence, Local; Transitional Cell, Carcinoma; Carcinoma in Situ; Mycobacterium
Keywords: Urinary Bladder Neoplasms; Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Urinary Bladder Diseases; Urologic Diseases; Mycobacterial cell wall DNA complex; Intravesical drug administration
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasm Recurrence, Local; Carcinoma, Transitional Cell; Carcinoma in Situ; Mycobacterium Infections; Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Urinary Bladder Diseases; Urologic Diseases | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EN3348 (Experimental): 8 mg mixed with sterile water for injection for a total volume of 50mL
  Interventions: Biological: EN3348
- Mitomycin C (Active Comparator): 40 mg powder will be reconstituted with sterile water for injection to a total volume of 40 mL
  Interventions: Biological: Mitomycin C

INTERVENTIONS:
Biological: EN3348 — Induction: 6 weekly instillations. Maintenance: Monthly instillations to Month 12
  Arms: EN3348
Biological: Mitomycin C — Induction: 6 weekly instillations. Maintenance: Monthly instillations to Month 12
  Arms: Mitomycin C

SUMMARY:
This is a phase 3 randomized, active-controlled, open-label, multicenter study that will be conducted in approximately 120 investigational sites worldwide. Subjects with either recurrent or refractory NMIBC (Ta high grade, T1 low or high grade, CIS) will be eligible for participation in this study.

Refractory disease is defined as evidence of persistent high grade bladder cancer (Ta HG, T1, and/or CIS) at least 6 months from the start of a full induction course of BCG with or without maintenance/re-treatment at 3 months.

Recurrent disease is defined as reappearance of disease after achieving a tumor-free status by 6 months following a full induction course of BCG with or without maintenance/re-treatment at 3 months. Subjects with recurrent disease must have recurred within 18 months following the last dose of BCG.

Approximately 450 subjects will be randomized. The primary objective of this study is to evaluate the efficacy of intravesical EN3348 as compared with mitomycin C in the treatment of subjects with recurrent or refractory NMIBC. The secondary objective is to evaluate the safety of EN3348 as compared with mitomycin C in the treatment of subjects with BCG recurrent or refractory NMIBC. This study will consist of 4 phases: Screening, Induction, Maintenance and Follow-Up and will be conducted over 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 years of age and older at time of consent signing
* Have either BCG recurrent or refractory NMIBC:

  * Refractory disease is defined as evidence of persistent high grade bladder cancer (Ta HG, T1 and/or CIS) at least 6 months from the start of a full induction course of BCG with or without maintenance/re-treatment at 3 months
  * Recurrent disease is defined as reappearance of disease after achieving a tumor-free status by 6 months following a full induction course of BCG with or without maintenance/re-treatment at 3 months. Subjects with recurrent disease must have recurred within 18 months following the last dose of BCG

    * A full induction course of BCG is defined as at least 5 out of 6 total expected instillations of BCG within a period of 2 months, regardless of dose strength
* Have histologically confirmed NMIBC (according to 2004 WHO classification) within 8 weeks prior to randomization

  * High grade Ta papillary lesion(s)
  * High or low grade T1 papillary lesion(s)(biopsy sample must include evidence of muscularis propria)
  * CIS, with or without Ta or T1 papillary tumor(s) of any grade
* Have had all visible papillary and resectable CIS lesion(s) removed by TURBT within 8 weeks prior to randomization
* Available for the duration of the study including follow-up (approximately 36 months)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status grade of 2 or less
* Have no evidence of urothelial carcinoma involving the upper urinary tract or the urethra (confirmed by extravesical work up, which may include radiological imaging and/or biopsy) within 6 months of randomization:

  * If previous work up occurred more than 6 months from randomization, extravesical work up must be repeated prior to randomization in order to determine eligibility
* Subjects (male and female) of child-bearing potential (including female subjects who are post-menopausal for less than 1 year) must be willing to practice effective contraception (as defined by the Investigator) during the study and be willing and able to continue contraception for 30 days after their last dose of study treatment
* Is able to understand and give written informed consent

Exclusion Criteria:

* Current or previous history of muscle invasive bladder tumors
* Current or previous history of lymph node positive and/or metastatic bladder cancer
* Current evidence of pure squamous cell carcinoma, pure adenocarcinoma or pure undifferentiated carcinoma of the bladder
* Currently receiving systemic cancer therapy (cytotoxic/cytostatic or immunotherapy)
* Currently receiving treatment with a prohibited therapy
* Current or prior history of systemic lupus erythematosus
* Systemic immunotherapy within 6 months of randomization
* Treatment with an investigational agent within 30 days or 5 half lives from randomization, whichever is longer
* Prior treatment with an intravesical chemotherapeutic agent within 3 months of randomization except for single perioperative dose of chemotherapy immediately post-TURBT
* Prior treatment with EN3348 (MCC) or any other mycobacterial cell wall composition or formulation
* Refractory to mitomycin C (failure to achieve tumor-free status following minimum of a 6 week induction course of mitomycin C)
* Contraindication to mitomycin C
* Untreated urinary tract or bladder infection
* ANC <1000/µL and hemoglobin <10 g/dL
* Known cardiovascular disease such as myocardial infarction within the past 3 months, unstable angina pectoris, congestive heart failure (NYHA Class III or IV) or uncontrolled cardiac arrhythmia
* Female subjects who are pregnant or lactating
* Congenital or acquired immune deficiency
* Have current or history of documented or suspected malignancy of any organ system (diagnosed, treated or untreated) within the past 5 years (with the exception of localized transitional cell carcinoma of the ureter treated with ureterectomy or nephroureterectomy, adequately treated basal cell or squamous cell carcinoma of the skin or asymptomatic non-metastatic prostate cancer either previously successfully treated or currently under active surveillance or receiving hormone therapy only)
* Bladder contracture or history of an inability to retain the instillate for a minimum of 1 hour, even with premedication
* Inability to tolerate intravesical administration or intravesical surgical manipulation (cystoscopy or biopsy)
* Clinically significant active infections
* Any medical or psychiatric condition which, in the opinion of the investigator, would preclude the participant from adhering to the protocol or completing the trial per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-11; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (72):
- United States (56):
  - Alaska Clinical Research Center, LLC, Anchorage, Alaska
  - BCG Oncology, PC, Phoenix, Arizona
  - Arizona Urologic Specialists, Tucson, Arizona
  - Urology Specialists of Southern California - Burbank, Burbank, California
  - Urology Specialist of Southern California - Encino, Encino, California
  - American Institute of Research, Los Angeles, California
  - San Diego Clinical Trials, San Diego, California
  - West Coast Clinical Research, Tarzana, California
  - Urology Specialists of Southern California - Torrance, Torrance, California
  - The Urology Center of Colorado, Denver, Colorado
  - Genitourinary Surgical Consultants, PC, Denver, Colorado
  - Urology Associates, Englewood, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Grove Hill Medical Center, New Britain, Connecticut
  - Florida Urological Associates, PA, Coral Springs, Florida
  - Urological Research Network, Hialeah, Florida
  - Urology Health Team, PLLC, Ocala, Florida
  - Advanced Research Institute, Inc., Trinity, Florida
  - Northwestern Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Northeast Indiana Research, LLC, Fort Wayne, Indiana
  - Kansas City Urology Care, P.A., Overland Park, Kansas
  - University of Maryland, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - Corbin Clinical Resources, Cumberland, Maryland
  - Chesapeake Urology Research Associates, Glen Burnie, Maryland
  - Myron I. Murdock, MD, LLC, Greenbelt, Maryland
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Bay State Urologists, Watertown, Massachusetts
  - Michigan Institute of Urology, Troy, Michigan
  - Delaware Valley Urology, LLC Burlington, Mount Laurel, New Jersey
  - Delaware Valley Urology, Voorhees Township, New Jersey
  - The Capital Region Medical Research Foundation, Inc., Albany, New York
  - Accumed Research Associates, Garden City, New York
  - Columbia University Medical Center, New York, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Montefiore Medical Center, The Bronx, New York
  - TriState Urologic Services PSC, Inc., Cincinnati, Ohio
  - Columbus Urology, Columbus, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Unison Clinical Research, Toledo, Ohio
  - Parkhurst Research Organization, LLC, Bethany, Oklahoma
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania
  - Urology Health Specialists, LLC, Bryn Mawr, Pennsylvania
  - Ilumina Clinical Associates, Indiana, Pennsylvania
  - Triangle Urological Group, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Mount Nittany Physician Group, State College, Pennsylvania
  - Pharma Resource, East Providence, Rhode Island
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Urology Associates of North Texas, Arlington, Texas
  - Urology Clinics of North Texas, PA, Dallas, Texas
  - Urology Associates of South Texas, McAllen, Texas
  - Virginia Urology, Richmond, Virginia
- Canada (9):
  - Southern Interior Medical Research, Inc., Kelowna, British Columbia
  - Pacific Urologic Research, Victoria, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Mor Urology Inc., Newmarket, Ontario
  - Office of Dr. Bernard Goldfarb, North Bay, Ontario
  - The Fe/Male Health Centres, Oakville, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital - University Health Network, Toronto, Ontario
  - Centre Hospitalier Universitaire de Quebec- L'Hotel-Dieu de Quebec, Québec, Quebec
- GUT (Society of Urologic Innovative Therapies), GbR, Kirchheim unter Teck, Germany
- Universitair Medisch Centrum St Radboud, Department of Urology, Nijmegen, Netherlands
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Oddział Urologii, Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie [Department of Urology, Independent Public Teaching Hospital #4 in Lublin], Lublin
  - Maria Sklodowska-Curie Institute of Oncology, Warsaw
  - Wojewódzki Szpital Specjalistyczny we Wrocławiu, Wroclaw
- Nottingham Urology Centre, NHS Trust, Nottingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- EN3348: 8 mg EN3348 mixed with water for injection for a total volume of 50mL
  EN3348: Induction: 6 weekly instillations. Maintenance: Monthly instillations to Month 12
- Mitomycin C: 40 mg mitomycin C mixed with water for injection to a total volume of 40 mL
  Mitomycin C: Induction: 6 weekly instillations. Maintenance: Monthly instillations to Month 12
Period: Overall Study
Arm/Group | EN3348 | Mitomycin C
Started | 39 | 45
Completed | 2 | 4
Not Completed | 37 | 41
Not completed — Study terminated early | 35 | 41
Not completed — Randomized but not treated | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EN3348 | Mitomycin C | Total
Number analyzed (Participants) | 39 | 45 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.0 (7.99) | 70.7 (11.18) | 71.8 (9.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 17
  Male | 34 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Event-free Survival of Intravesical EN3348 With Mitomycin C.
Description: Primary efficacy endpoint will be event-free survival - the interval from randomization to an event. An event is defined as tumor recurrence, tumor progression to muscle invasive bladder cancer or death, whichever occurs first. Tumor recurrence or progression must be documented by bladder biopsy.
Time Frame: 1 year
Population: The study was discontinued early. The number of subjects randomized at time of closure represented 18.7% of the planned enrollment of 450 subjects. Thus, the planned analysis as stated in the protocol was not performed. Only 2 subjects (5.1%) in the EN3348 arm and 4 subjects (8.9%) in the mitomycin C arm completed all planned doses.
Groups:
- EN3348: 8 mg mixed with water for injection for a total volume of 50mL
  Treatment - Induction (6 weekly instillations) followed Maintenance (monthly instillations up to Month 12)
- Mitomycin C: 40 mg mixed with water for injection to a total volume of 40 mL
  Treatment - Induction (6 weekly instillations) followed Maintenance (monthly instillations up to Month 12)
Arm/Group | EN3348 | Mitomycin C
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Comparison of Safety of EN3348 With Mitomycin C [Adverse Events (Other Than Serious Adverse Events) With Frequency Threshold of 5% or Greater].
Description: Safety endpoint displayed includes adverse events (other than serious adverse events) with a frequency threshold of 5% or greater, for each treatment arm. No statistical comparisons have been performed between the 2 treatment arms.
Time Frame: Through study early termination, approximately 23 months from first subject enrolled.
Population: Relevant safety data are presented in the Adverse Events and Serious Adverse Events Modules. Any clinically significant findings pertaining to other secondary outcomes such as vital signs, physical exams and laboratory test results would appear in these Modules as well. No statistical comparisons have been performed between the 2 treatment arms.
Measure: Number; unit: participants
Groups:
- EN3348: 8 mg mixed with sterile water for injection for a total volume of 50mL
  Treatment - Induction (6 weekly instillations) followed by Maintenance (monthly instillations up to Month 12)
- Mitomycin C: 40 mg mixed with sterile water for injection to a total volume of 40 mL
  Treatment - Induction (6 weekly instillations) followed by Maintenance (monthly instillations up to Month 12)
Arm/Group | EN3348 | Mitomycin C
Number analyzed (Participants) | 37 | 45
participants
  Dysuria | 9 | 12
  Hematuria | 7 | 3
  Pollakiuria | 6 | 6
  Fatigue | 6 | 3
  Urinary tract infection | 5 | 5
  Diarrhea | 3 | 2
  Back pain | 2 | 4
  Nausea | 2 | 3

ADVERSE EVENTS:
Arm/Group | EN3348 | Mitomycin C
Serious Adverse Events (participants affected / at risk) | 4/37 | 2/45
Other Adverse Events (participants affected / at risk) | 32/37 | 35/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EN3348 (N=37) | Mitomycin C (N=45)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bladder spasms (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 1 (1) | 0 (0)
Post-procedural hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EN3348 (N=37) | Mitomycin C (N=45)
Dysuria (Renal and urinary disorders) | 9 | 12
Hematuria (Renal and urinary disorders) | 7 | 3
Pollakiuria (Renal and urinary disorders) | 6 | 6
Diarrhea (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 3
Fatigue (General disorders) | 6 | 3
Urinary tract infection (Infections and infestations) | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other